CLINICAL TRIAL: NCT07338981
Title: (CHRONO-RCC) Time-of-day-Dependent Administration of Dual Immune Check Point Inhibitors (ICI) in Advanced Kidney Cancer
Brief Title: The Impact of Time-of-day-Dependent Administration of Nivolumab-Ipilimumab (ICI/ICI) Combination on Overall Survival in Adults With Advanced Kidney Cancer: A Pragmatic Multicenter, Randomized Controlled Trial.
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Guliz Ozgun (Other)
Collaborators: British Columbia Cancer Agency (Other)
Responsible Party: Sponsor-Investigator, Guliz Ozgun, Medical Oncologist, Principal Investigator, British Columbia Cancer Agency
Organization: British Columbia Cancer Agency (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Chrono-RCC
Record Dates: First submitted 2025-12-05; First posted 2026-01-14 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Advanced Kidney Cancer
Keywords: Chronoimmunotherapy; Time-of-day administration; Chronotherapy; Circadian rhythm; Advanced kidney cancer; Nivolumab/Ipilimumab
MeSH Terms: interventions — Nivolumab; Ipilimumab

STUDY DESIGN:
Intervention Model Description: This study is a randomized, controlled trial designed to evaluate the effects of timing of standard-of-care (SOC) treatment administration on patient outcomes. Participants will be randomly assigned to receive SOC nivolumab/ipilimumab either in the morning or in the afternoon, with no additional interventions planned. Patients will be scheduled for treatments at the same time for the first four cycles, with a ±1 hour flexibility, to minimize the impact of timing as a confounding factor in the analyses. The trial is open-label and not blinded due to the nature of the intervention (timing of treatment).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm A: Morning ICI/ICI Treatment (Active Comparator): Participants will receive standard-of-care therapy (ICI/ICI) administered in the morning (before 11:30am).
  Interventions: Drug: Nivolumab & Ipilimumab
- Arm B: Afternoon ICI/ICI Treatment (Active Comparator): Participants will receive standard-of-care therapy (ICI/ICI) administered in the afternoon (after 1:30pm).
  Interventions: Drug: Nivolumab + Ipilimumab

INTERVENTIONS:
Drug: Nivolumab & Ipilimumab — Participants will receive ICI/ICI as part of their standard-of-care therapy administered in the morning before 11:30am (Arm A) , as determined by randomization.
  Other Names: ICI/ICI
  Arms: Arm A: Morning ICI/ICI Treatment
Drug: Nivolumab + Ipilimumab — Participants will receive ICI/ICI as part of their standard-of-care therapy administered in the afternoon after 1:30pm (Arm B) , as determined by randomization.
  Arms: Arm B: Afternoon ICI/ICI Treatment

SUMMARY:
The goal of this clinical trial is to learn if the timing of treatments plays a role in how effective the standard-of-care drugs nivolumab/ipilimumab (ICI/ICI) works to treat adults with advanced kidney cancer. The trial will also learn if time-of-day reduces ICI/ICI side-effects. Researchers will compare ICI/ICI given in the morning (before 11:30am) vs in the afternoon (after 1:30pm), to see if circadian rhythm effects how ICI/ICI works to treat advanced kidney cancer. Participants will be randomized in Arm A or Arm B to receive drugs ICI/ICI either in the morning (Arm A) or afternoon (Arm B) as part of their standard-of-care treatment for advanced kidney cancer. Participants will:

* Visit the clinic either in the morning (Arm A) or afternoon (Arm B) to receive ICI/ICI treatment as part of their regular medical care for advanced kidney cancer
* Frequency of visits will follow standard-of-care guidelines

ELIGIBILITY:
Inclusion Criteria:

Participants must meet all of the following criteria to be eligible for participation in this trial. Waivers to the inclusion criteria will NOT be allowed.

1. Age 18 or older
2. Able to provide informed consent
3. Histologically confirmed advanced clear cell kidney cancer
4. Eligible for standard-of-care nivolumab/ipilimumab regimen
5. Measurable disease per RECIST 1.1
6. ECOG performance status 0-2
7. Ability to adhere to scheduled infusion times (Before 11:30 a.m. or after 1:30 pm)

Exclusion Criteria:

Participants are excluded from the trial if any of the following criteria apply. Waivers to the exclusion criteria will NOT be allowed.

1. Non-clear cell RCC histology
2. Concurrent malignancy requiring active systemic therapy, unless disease-free for at least 2 years
3. Inability to comply with protocol-specified infusion timing for the first 4 cycles
4. Night shift workers
5. Clinical evidence of new or enlarging brain metastasis or carcinomatous meningitis
6. Known psychiatric or substance abuse disorder that would interfere with cooperation with the requirements of the trial
7. Patients who have traveled across ≥2 time zones within the past 14 days prior to randomization will be excluded, due to potential disruption of circadian rhythms (jet lag), which may affect chronotherapy-related endpoints.
8. Patients with a clinically diagnosed sleep disorder, including but not limited to insomnia, obstructive sleep apnea, restless leg syndrome, or circadian rhythm sleep-wake disorders, that is moderate to severe, untreated, or poorly controlled, will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Estimated)
Dates: Start 2026-04 (Estimated); Primary Completion 2030-12 (Estimated); Study Completion 2032-12 (Estimated)

PRIMARY OUTCOMES:
Assess Overall-Survival in time-of-day administration of ICI/ICI treatment | From enrollment to the end of follow-up at 24 months.
  To assess overall survival (OS) in patients treated with time-of day dependent administration of nivolumab-ipilimumab (ICI/ICI) standard-of-care therapy in advanced kidney cancer. OS is defined as the time from randomization to death from any cause. The primary analysis will compare OS curves between study arms and estimate 2-year OS rates for each group.

SECONDARY OUTCOMES:
Determine Objective Response Rate in time-of-day administration of ICI/ICI treatment | From enrollment to the end of follow-up at 24-months.
  Objective response rate (ORR) will be determined by Proportion of patients achieving a complete or partial response as assessed by RECIST v1.1 criteria, confirmed by central or investigator review. Tumor assessments will be performed as standard of care (typically every 12 weeks), and best overall response prior to disease progression will be used for ORR determination.
Evaluate Progression-Free Survival in time-of-day administration of ICI/ICI treatment | From enrollment to the end of follow-up at 24-months.
  Progression-free Survival (PFS) will be determined by time of randomization to disease progression or death from any cause.
Determine the Time-to-Treatment Failure in time-of-day administration of ICI/ICI treatment | From enrollment to the end of follow-up at 24-months.
  Time to treatment failure (TTF) is determined by assessing time from treatment initiation to treatment discontinuation for any reason, including disease progression, unacceptable toxicity, patient withdrawal, or death, capturing both treatment efficacy and tolerability.
Assess treatment-related tolerability and toxicity differences | From enrollment to the end of follow-up at 24-months.
  Differences in steroid use (yes/no) for the management of treatment-related toxicity, treatment interruptions (yes/no) due to treatment-related toxicity, and treatment discontinuations (yes/no) due to treatment-related toxicity will be used as surrogate safety outcomes, as comprehensive adverse event documentation is beyond the scope of this pragmatic clinical trial. The study seeks to determine whether treatment administration at a predefined time of day is associated with differences in the need for toxicity-related clinical interventions. Given that the relevant adverse events are well characterized in the existing literature, the focus of this study is on comparative safety between groups using these surrogate measures rather than on detailed characterization of individual adverse events.
Immune Profiling | At 4 time points: Baseline, 1-day post first cycle of treatment, 3 weeks into treatment and 12 weeks into treatment
  Immune cell populations will be characterized from the blood samples at baseline (prior to treatment initiation) and at three predefined time points during therapy: 1 day after treatment initiation, 3 weeks into treatment, and 12 weeks into treatment. Cytometry by time-of-flight (CyTOF) will be used to comprehensively profile immune cell populations allowing for high-dimensional assessment of immune cell composition and activation states across treatment timing groups.
Bulk RNA sequencing (RNA-seq) | At 4 time points: Baseline, 1-day post first cycle of treatment, 3 weeks into treatment and 12 weeks into treatment
  Bulk RNA sequencing (RNA-seq) will be performed to comprehensively characterize global gene expression profiles and to evaluate time-of-day-associated differences in immune-related transcriptional signatures. This approach will enable the identification of circadian variation in gene expression and provide insight into temporal regulation of immune pathways in response to treatment.
Cytokine and chemokine analyses | At 4 time points: Baseline, 1-day post first cycle of treatment, 3 weeks into treatment and 12 weeks into treatment
  Plasma will be isolated for cytokine and chemokine analyses to assess systemic immune signaling and inflammatory profiles. Quantitative evaluation of circulating cytokines and chemokines will provide insight into treatment- and time-dependent changes in immune activation, inflammation, and immune regulation, complementing cellular and transcriptional immune profiling.

CONTACTS AND LOCATIONS:
Locations (1):
- BC Cancer - Vancouver Cancer Centre, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Wang C, Zeng Q, Gul ZM, Wang S, Pick R, Cheng P, Bill R, Wu Y, Naulaerts S, Barnoud C, Hsueh PC, Moller SH, Cenerenti M, Sun M, Su Z, Jemelin S, Petrenko V, Dibner C, Hugues S, Jandus C, Li Z, Michielin O, Ho PC, Garg AD, Simonetta F, Pittet MJ, Scheiermann C. Circadian tumor infiltration and function of CD8+ T cells dictate immunotherapy efficacy. Cell. 2024 May 23;187(11):2690-2702.e17. doi: 10.1016/j.cell.2024.04.015. Epub 2024 May 8. PMID 38723627
- [Background] Fortin BM, Pfeiffer SM, Insua-Rodriguez J, Alshetaiwi H, Moshensky A, Song WA, Mahieu AL, Chun SK, Lewis AN, Hsu A, Adam I, Eng OS, Pannunzio NR, Seldin MM, Marazzi I, Marangoni F, Lawson DA, Kessenbrock K, Masri S. Circadian control of tumor immunosuppression affects efficacy of immune checkpoint blockade. Nat Immunol. 2024 Jul;25(7):1257-1269. doi: 10.1038/s41590-024-01859-0. Epub 2024 May 28. PMID 38806707
- [Background] Lee Y. Roles of circadian clocks in cancer pathogenesis and treatment. Exp Mol Med. 2021 Oct;53(10):1529-1538. doi: 10.1038/s12276-021-00681-0. Epub 2021 Oct 7. PMID 34615982
- [Background] Karaboue A, Innominato PF, Wreglesworth NI, Duchemann B, Adam R, Levi FA. Why does circadian timing of administration matter for immune checkpoint inhibitors' efficacy? Br J Cancer. 2024 Sep;131(5):783-796. doi: 10.1038/s41416-024-02704-9. Epub 2024 Jun 4. PMID 38834742
- [Background] Dizman N, Govindarajan A, Zengin ZB, Meza L, Tripathi N, Sayegh N, Castro DV, Chan EH, Lee KO, Prajapati S, Feng M, Loo V, Pace M, O'Brien S, Bailey E, Barragan-Carrillo R, Chehrazi-Raffle A, Hsu J, Li X, Agarwal N, Pal SK. Association Between Time-of-Day of Immune Checkpoint Blockade Administration and Outcomes in Metastatic Renal Cell Carcinoma. Clin Genitourin Cancer. 2023 Oct;21(5):530-536. doi: 10.1016/j.clgc.2023.06.004. Epub 2023 Jun 25. PMID 37495481
- [Background] Patel JS, Woo Y, Draper A, Jansen CS, Carlisle JW, Innominato PF, Levi FA, Dhabaan L, Master VA, Bilen MA, Khan MK, Lowe MC, Kissick H, Buchwald ZS, Qian DC. Impact of immunotherapy time-of-day infusion on survival and immunologic correlates in patients with metastatic renal cell carcinoma: a multicenter cohort analysis. J Immunother Cancer. 2024 Mar 26;12(3):e008011. doi: 10.1136/jitc-2023-008011. PMID 38531662
- [Background] Giacchetti S, Bjarnason G, Garufi C, Genet D, Iacobelli S, Tampellini M, Smaaland R, Focan C, Coudert B, Humblet Y, Canon JL, Adenis A, Lo Re G, Carvalho C, Schueller J, Anciaux N, Lentz MA, Baron B, Gorlia T, Levi F; European Organisation for Research and Treatment of Cancer Chronotherapy Group. Phase III trial comparing 4-day chronomodulated therapy versus 2-day conventional delivery of fluorouracil, leucovorin, and oxaliplatin as first-line chemotherapy of metastatic colorectal cancer: the European Organisation for Research and Treatment of Cancer Chronotherapy Group. J Clin Oncol. 2006 Aug 1;24(22):3562-9. doi: 10.1200/JCO.2006.06.1440. PMID 16877722
- [Background] Levi F, Okyar A, Dulong S, Innominato PF, Clairambault J. Circadian timing in cancer treatments. Annu Rev Pharmacol Toxicol. 2010;50:377-421. doi: 10.1146/annurev.pharmtox.48.113006.094626. PMID 20055686
- [Background] Motzer RJ, Tannir NM, McDermott DF, Aren Frontera O, Melichar B, Choueiri TK, Plimack ER, Barthelemy P, Porta C, George S, Powles T, Donskov F, Neiman V, Kollmannsberger CK, Salman P, Gurney H, Hawkins R, Ravaud A, Grimm MO, Bracarda S, Barrios CH, Tomita Y, Castellano D, Rini BI, Chen AC, Mekan S, McHenry MB, Wind-Rotolo M, Doan J, Sharma P, Hammers HJ, Escudier B; CheckMate 214 Investigators. Nivolumab plus Ipilimumab versus Sunitinib in Advanced Renal-Cell Carcinoma. N Engl J Med. 2018 Apr 5;378(14):1277-1290. doi: 10.1056/NEJMoa1712126. Epub 2018 Mar 21. PMID 29562145